CLINICAL TRIAL: NCT04945070
Title: INSULIN THERAPY DE-INTENSIFICATION WITH iGlarLixi
Acronym: IDEAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Martin Haluzik, prof. MUDr. Martin Haluzik, DrSc., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEAL V2.2
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iGlarLixi (Experimental): Subjects switched from MDI to iGlarLixi
  Interventions: Drug: IGlarLixi
- Control (Active Comparator): Patients continuing with previous MDI
  Interventions: Drug: MDI - Multiple dose insulin injection

INTERVENTIONS:
Drug: IGlarLixi — Switching T2DM subjects from MDI to iGlarLixi
  Arms: iGlarLixi
Drug: MDI - Multiple dose insulin injection — Continuing with established MDI regimen
  Arms: Control

SUMMARY:
Intensive insulin therapy using multiple daily injections (MDI) constitutes the most intense type of regimen in type 2 diabetes mellitus (T2D). Although highly effective in lowering blood glucose, it can also increase the risk of hypoglycemia, promote weight gain and cause significant treatment burden for the patients. As demonstrated by a number of clinical studies, overtreatment is a common and generally unrecognized problem in patients with T2D; nevertheless, medication de-escalation is still infrequent in everyday clinical practice. IGlarLixi is a once-daily fixed-ratio combination (FRC) of a basal insulin and a glucagon-like peptide-1 receptor agonist (GLP-1 RA), which can offer similar efficacy in glucose control with lower rates of hypoglycemia and smaller weight gain that basal insulin regimens. The aim of our randomised, controlled study is to examine prospectively the safety and efficacy of de-escalating MDI regimens to iGlarLixi in T2D adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Adult participants with T2DM
* Participants who have been treated with a an MDI regimen comprising of at least 3 doses of prandial insulin per day and one dose of basal insulin per day for at least 3 months before the screening visit,
* Participants treated with metformin (unless intolerance to metformin use is present) ± SGLT2i at stable doses for at least 3 months prior screening.
* Total daily insulin dose ≤ 0.8 IU/kg,
* Fasting C peptide above the lower limit of the normal range,
* HbA1c at screening visit ≤ 75 mmol/mol (9%) as measured by local laboratory,
* HbA1c at screening visit 76-86 mmol/mol (9.1-10%) as measured by local laboratory in case of proven non-compliance with MDI regimen

Exclusion Criteria:

* At screening visit, age under legal age of adulthood (<18 years),
* History of other diabetes than T2DM (type 1 diabetes T1DM, monogenic, secondary..)
* Use of any oral or injectable glucose-lowering agents other than those stated in the inclusion criteria within the last 3 months before screening,
* History of discontinuation of a previous treatment with GLP-1 RA for safety/tolerability reasons or lack of efficacy,
* Use of systemic glucocorticoids (excluding topical and inhaled forms) for a total duration of 1 week or more within 3 months prior to screening visit,
* Comorbidity (such as but not limited to rheumatoid arthritis) with continuous, intermittent or expected systemic glucocorticoid therapy during the next 30 weeks after screening visit,
* Use of weight loss drugs within 3 months prior to screening visit,
* Use of any investigational drug within 1 month or 5 half-lives, whichever is longer, prior to screening visit,
* Within the last 3 months prior to screening visit: history of stroke, pulmonary embolism, myocardial infarction, unstable angina, or heart failure requiring hospitalization,
* Chronic hear failure NYHA stages III-IV
* Acute or chronic liver failure - established diagnosis of acute or chronic liver failure (Child-Pugh 3, MELD≥15) or liver cirrhosis
* Planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period,
* Known history of drug or alcohol abuse within 6 months prior to the time of screening visit,
* Active malignancy
* Anaemia with haemoglobin < 100 g/l at baseline
* Participants with conditions/concomitant diseases making them non evaluable for the efficacy endpoints (eg, hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within the last 3 months prior to the screening visit),
* Participants with conditions/concomitant diseases precluding their safe participation in this study (eg, active malignant tumor, major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require treatment within the study period, etc.),
* Impossibility to meet specific protocol requirements (eg, scheduled visits, participants unable to fully understand participant's study documents and to complete them, etc.),
* Uncooperative or any condition that could make the participant potentially non-compliant to the study procedures (eg, participant unable or unwilling to do self-injections or blood glucose monitoring using the sponsor-provided blood glucose meter at home, etc.);
* Participant is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Participation in another clinical trial
* Pregnancy or lactation,
* Women of childbearing potential not protected by highly effective contraceptive method of birth control (definition see section 10.1.1.1),
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (ie, worsening) or not controlled (ie, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening visit or history of surgery affecting gastric emptying
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy had now been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy,
* Personal or immediate family history of MTC or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia syndromes),
* Participant who has a renal function impairment with creatinine clearance <30 mL/min (using the eGFR) or end-stage renal disease (ie. CKD stage IV or V),
* History of allergic reaction to any GLP-1 RA in the past

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 6 months
  The effect of the transition from MDI regimen to IGlarLixi on HbA1c values

SECONDARY OUTCOMES:
Hypoglycemia | 6 months
  Number and time in hypoglycemia
Compliance | 6 months
  Adherence to treatment and recommended SMBG pattern
Fasting plasma glucose | 6 months
Postprandial plasma glucose | 6 months
Glycemic variability | 6 months
  Measured from continuous glucose monitoring
Time in target range of 3.9-10 mmol/l | 6 months
  Measured from continuous glucose monitoring
Body weight | 6 months
  Change in body weight
Treatment Satisfaction | 6 months
  Assessment of quality of life using Diabetes Treatment Satisfaction Questionnaire

OTHER OUTCOMES:
ALT | 6 months
  Marker of hepatic steatosis
hsCRP | 6 months
  Marker of low-grade inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Novodvorsky P, Thieme L, Lankova I, Mraz M, Taybani ZJ, Botyik B, Stella P, Vytasil M, Lauand F, Bonnemaire M, Haluzik M. The IDEAL (Insulin therapy DE-intensificAtion with iglarLixi) Randomised Controlled Trial-Study Design and Protocol. Diabetes Ther. 2024 Jun;15(6):1461-1471. doi: 10.1007/s13300-024-01582-x. Epub 2024 Apr 24. PMID 38653903